CLINICAL TRIAL: NCT04168307
Title: Conventional Physiotherapy Versus Use of a New Ankle Trainer Device After Weber b Ankle Fracture Operation. A Randomized Controlled Trial
Brief Title: Physiotherapy Versus Use of a New Ankle Trainer Device After Ankle Fracture Operation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marius Molund, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUN studien
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Ankle Fracture - Lateral Malleolus; Post-Op Complication
Keywords: ankle fracture; rehabilitation
MeSH Terms: conditions — Ankle Fractures; Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The physiotherapist conducting follow ups at 6, 12 and 52 weeks was masked for group affiliation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankle trainer device (Experimental): The patients were instructed in the use of a new spring loaded ankle trainer
  Interventions: Device: Ankle trainer device
- Conventional physiotherapy (Active Comparator): The patients were instructed in passive stretching exercises by the use of a non-elastic band
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: Ankle trainer device — The ankle trainer provides passive stretch in dorsal flexion of the ankle as well as active plantar flexion.
  Arms: Ankle trainer device
Other: Conventional physiotherapy — The patients were instructed in stretching exercises using a non-elastic band
  Arms: Conventional physiotherapy

SUMMARY:
The study will compare the functions outcomes between two different rehabilitation protocol after operated weber b ankle fractures

DETAILED DESCRIPTION:
Patients that are operated for weber b ankle fractures will after the surgery be randomized into two different post operative rehabilitation protocols. One group will receive conventional physiotherapy with stretching of the ankle with a non-elastic band, while the other group will use a new spring-loaded ankle trainer. The rehabilitation will continue for 3 weeks. Patients will be evaluated with the Olerud Molander ankle score and visual analog scale for pain at 3, 6, 12 and 52 weeks follow-up. Length of hospitalization and all adverse events will be registered. Ankle range of motion will be registered at 6, 12 and 52 weeks

ELIGIBILITY:
Inclusion Criteria:

* Weber b ankle fracture. Exercise stable osteosynthesis. Good compliance

Exclusion Criteria:

* Previous trauma to the tibia or fibula. Previous ankle or foot surgery. Sympthomatic arthritis or generalized joint disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-11-29 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Olerud Molander ankle score (OMAS) | 52 weeks after surgery
  A patient related outcome measure that evaluates ankle function on a 0-100 scale. 100 is indicating a perfect result

SECONDARY OUTCOMES:
Visual analog scale for pain (VAS) | 52 weeks
  Describes pain on a 0-10 scale with 0 representing no pain, and 10 the worst imaginable pain
Ankle range of motion | 52 weeks
  Ankle dorsiflexion measured am Lindsjø

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, MD, Principal Investigator — Oslo University Hospital

IPD SHARING:
Plan to Share IPD: No
There is no such plan